CLINICAL TRIAL: NCT03109314
Title: The Effect of Donepezil on Perceptual Learning in Adult Amblyopia
Brief Title: Combining Donepezil With Perceptual Learning in Normal and Amblyopic Human The Effect of Donepezil on Perceptual Learning in Adult Amblyopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dennis Levi (Other)
Responsible Party: Sponsor-Investigator, Dennis Levi, Professor of Optometry and Vision Science, University of California, Berkeley
Organization: University of California, Berkeley (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 020976_01
Record Dates: First submitted 2017-03-23; First posted 2017-04-12 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Amblyopia
Keywords: amblyopia; donepezil; perceptual learning; crowding; contrast sensitivity; visual acuity
MeSH Terms: conditions — Amblyopia; Crowding | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single-letter training group (Active Comparator): Subjects will be trained on a low-contrast single-letter task. The task is to identify a faint letter (low-contrast). Performance will be measured as correct or incorrect. Training will consist of identifying these low-contrast letters for 1000 trials per day (10 blocks of 100 trials each, subjects can take breaks in-between blocks), for a total of 10 days. During training, subjects will be administered a daily dosage of 5 mg of donepezil. Immediately before and after training (the day before and the day after), subjects' performance on (1) visual acuity; (2) contrast for identifying letters and (3) crowding extent will be measured.
  Interventions: Drug: Donepezil; Behavioral: Single-letter training
- Uncrowd training group (Active Comparator): Subjects will be trained on an uncrowd task (identifying the middle letter of groups of three letters presented). Performance will be measured as correct or incorrect. Training will consist of identifying these letters for 1000 trials per day (10 blocks of 100 trials each, subjects can take breaks in-between blocks), for a total of 10 days. During training, subjects will be administered a daily dosage of 5 mg of donepezil. Immediately before and after training (the day before and the day after), subjects' performance on (1) visual acuity; (2) contrast for identifying letters and (3) crowding extent will be measured.
  Interventions: Drug: Donepezil; Behavioral: Uncrowd training

INTERVENTIONS:
Drug: Donepezil — Donepezil will be administered to subjects three days before each training, and during training, to evaluate if donepezil improves the effectiveness of training.
  Other Names: Aricept
Behavioral: Single-letter training — Subjects will undergo training to identify single letters (10,000 trials, or 10 blocks per session for 10 sessions).
  Arms: Single-letter training group
Behavioral: Uncrowd training — Subjects will undergo training to identify letters closely flanked by other letters (10,000 trials, or 10 blocks per session for 10 sessions).
  Arms: Uncrowd training group

SUMMARY:
The research deals with amblyopia or lazy eye, a condition that affects about 3% of the population, and results in a variety of visual deficits. Recent work suggests that there is limited neural plasticity in the visual system of adults with amblyopia. This study is aimed at understanding and increasing this plasticity. In this study, the investigators aim to understand how the amblyopic brain learns and how this process is affected by a drug called donepezil, which is sometimes given as a treatment for Alzheimer's disease. The investigators hope that this study will help to identify the chemical components that help the brain to learn, as well as the mechanism of amblyopia. The investigators also plan to test the normal periphery, as control.

DETAILED DESCRIPTION:
The research deals with amblyopia or lazy eye, a condition that affects about 3% of the population, and results in a variety of visual deficits. Recent work suggests that there is limited neural plasticity in the visual system of adults with amblyopia. This study is aimed at understanding and increasing this plasticity. In this study, the investigators aim to understand how the amblyopic brain learns and how this process is affected by a drug called donepezil, which is sometimes given as a treatment for Alzheimer's disease. The investigators hope that this study will help to identify the chemical components that help the brain to learn, as well as the mechanism of amblyopia. The investigators also plan to test the normal periphery, as control.

In this study, donepezil will be administered while amblyopic subjects (or normally sighted subjects tested in the periphery) are trained on a low-contrast single-letter recognition task, or an uncrowd task (recognizing a letter closely embedded within two other letters). Subjects will be asked to identify the target letter (the low-contrast single letter, or the letter embedded within other letters). Training will take place for 10 consecutive days. Pre- and post-tests will be conducted immediately before and after training, and will consist of the measurements of visual acuity, crowding extent and contrast threshold for recognizing single letters.

ELIGIBILITY:
Subjects with amblyopia

Inclusion Criteria:

* corrected visual acuity being 20/30 or worse in the poorer eye (at least 20/20 in the better eye)
* reduced stereoacuity
* normal retina

Exclusion Criteria:

* with other diagnosed eye diseases

Subjects with normal vision

Inclusion Criteria:

* corrected visual acuity at least 20/20 in each eye
* normal stereoacuity
* normal retina

Exclusion Criteria:

* with other diagnosed eye diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement in percent-correct performance in the respective training task | During training (performance will be summarized for each block of trials (a block takes approximately 5 - 10 min to complete). In other words, there should be 100 points of measurements throughout the training period.)
  During training, for each trial, participants' responses can be categorized as correct or incorrect. The investigators will use the percent-correct performance to quantify the performance in each block, and this percent-correct performance will be measured throughout training (i.e. for each block on each day (10 blocks per day), and for 10 training days).
Visual acuity (the smallest letter the participants can see) | Immediately (one day) before and after training
  The change in visual acuity before and after (one day before and one day after) training will be compared. The change will be expressed as a ratio.
Contrast sensitivity for identifying single letters (the lowest contrast required to identify letters) | Immediately (one day) before and after training
  Contrast refers to the smallest difference in luminance between a letter and its background. This is a standard clinical measurement. Essentially, the lowest contrast letter is also the faintest letter that a participant can see. The change in contrast sensitivity for identifying single letters before and after (one day before and one day after) training will be compared. The change will be expressed as a ratio.
Crowding extent (the extent over which adjacent letters will affect the recognition of a letter) | Immediately (one day) before and after training
  Crowding extent refers to the minimum distance between adjacent letters such that the presence of adjacent letters affects the recognition of a target letter. Usually the letter separation will be adjusted until the adjacent letters no longer affects how well the middle letter can be recognized. This distance is the crowding extent. The change in the crowding extent before and after (one day before and one day after) training will be measured. The change will be expressed as a ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Levi, OD, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chung STL, Li RW, Silver MA, Levi DM. Donepezil Does Not Enhance Perceptual Learning in Adults with Amblyopia: A Pilot Study. Front Neurosci. 2017 Aug 7;11:448. doi: 10.3389/fnins.2017.00448. eCollection 2017. PMID 28824369
- See also: Article in Frontiers in Neuroscience — https://www.frontiersin.org/articles/10.3389/fnins.2017.00448/full